CLINICAL TRIAL: NCT03182998
Title: Testing Decision Aids to Improve Prostate Cancer Decisions for Minority Men
Brief Title: Decision Aids to Improve Knowledge in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jon C. Tilburt, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-010459; R01MD008934-05 (NIH)
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Knowing Your Options) (Experimental): Arm A ("Knowing your Options") Patients receive "Knowing your Options" decision aid before their consultation visit.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis
- Arm B (Prostate Choice) (Experimental): Patients receive "Prostate Choice" decision aid during their consultation visit.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis
- Arm C (Usual Care) (Active Comparator): Patients undergo usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Internet-Based Intervention — Receive "Knowing your Options" decision aid
  Arms: Arm A (Knowing Your Options)
Other: Internet-Based Intervention — Receive "Prostate Choice" decision aid
  Arms: Arm B (Prostate Choice)
Other: Best Practice — Undergo usual care
  Other Names: best practice, Best Practice, standard of care, standard therapy
  Arms: Arm C (Usual Care)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment, Quality-of-Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase III trial studies how well decision aids work in improving knowledge in patients with prostate cancer. Decision aids may improve patients' knowledge of their condition and options for treatment, and may also help when talking with their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have prostate biopsy within 4 months prior to registration showing newly diagnosed prostate cancer, stage T1-3N0M0; in addition, patients must have: Gleason score 6-10
* Prostate-specific antigen (PSA) < 50 ng/mL
* Patients who have had a history of non-cutaneous malignancy in the previous 5 years are not eligible; exception: patients with history of non-melanoma skin cancer are eligible
* Scheduled prostate cancer consultation to be the first consultation after diagnosis (i.e. not a second-opinion or a consultation following previous discussions of treatment options)
* Patients may not be concurrently enrolled to another clinical trial for the treatment of cancer; co-enrollment to biospecimen studies is allowed
* Patients with impaired decision-making capacity (such as with a diagnosis of dementia or memory loss) are not eligible for this study
* Patients must be able to read and comprehend English; non-English-speaking patients may participate so long as an interpreter (e.g., family member, clinic staff, etc.) is present for consent, for the decision aid administration, and gathering of baseline and follow-up measures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon C. Tilburt, M.D., Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Alaska Native Tribal Health Consortium, Anchorage, Alaska
  - Mayo Clinic, Scottsdale, Arizona
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Metrohealth Medical Center Urology Institute, Cleveland, Ohio
  - Regional Health, Rapid City, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care)
Started | 37 | 33 | 33
Completed | 36 | 33 | 33
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care) | Total
Number analyzed (Participants) | 37 | 33 | 33 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.49 (6.57) | 65.16 (6.25) | 64.52 (8.07) | 64.34 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 37 | 33 | 33 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 35 | 30 | 31 | 96
  Unknown or Not Reported | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 6 | 17
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 5 | 4 | 16
  White | 24 | 22 | 23 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 33 | 33 | 103
Treatment Preferred [Count of Participants; unit: Participants]
  Surgery | 15 | 13 | 16 | 44
  Radiation | 9 | 6 | 8 | 23
  Active surveillance | 5 | 4 | 4 | 13
  Unsure | 6 | 10 | 5 | 21
  Missing | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Assessed by Prostate Cancer Treatment Questionnaire
Description: The primary outcome, knowledge, will be assessed by a standardized questionnaire (i.e., Prostate Cancer Treatment Questionnaire) administered once, immediately after the clinical consultation while the patient is still at the study site. The number correct from this 12-item measure will be reduced to a proportion of total number correct. With 1.0 (12 out of 12 item average) being the best possible outcome and 0.0 (0 out of 12 item average) the worst possible outcome
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care)
Number analyzed (Participants) | 36 | 33 | 33
score on a scale | 0.69 (0.16) | 0.69 (0.18) | 0.64 (0.20)

2. Secondary Outcome: Decisional Quality as Measured by Decisional Regret Scale
Description: The Decisional Regret Scale is a short, 5-item scale measuring "distress or remorse after a (health care) decision." The instrument has been validated in other decision aid studies. Questions are answered on a 5-point agreement scale. A score of 0 means no decisional regret and 5 is the maximum level of regret. The continuous scores were then grouped into two categories, 0 (no regret) and 1+ (at least some regret).
Time Frame: 12 months
Population: Secondary outcomes were to be based on data collected at 12 months. Two of our sites (enrolling >50% of study participants) experienced staff turnover and/or loss of contact with participants. As a result, we lost our ability and opportunity to maintain contact with nearly all participants at both sites and were unable to collect secondary outcome data at 12 months. Results reported here reflect the data we were able to collect.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care)
Number analyzed (Participants) | 5 | 5 | 7
Participants
  Decisional Regret Total score of 0 | 2 | 3 | 2
  Decisional Regret Total score of 1+ | 3 | 2 | 5

3. Secondary Outcome: Quality of Life Assessed by Questionnaire
Description: The Expanded Prostate Cancer Index Composit (EPIC-26) measures health-related quality of life and returns summary scores for urinary, bowel, sexual, and hormonal domains with high test-retest reliability and internal consistency. Scores will be converted into continuous summary scores using standard algorithms. For the EPIC-26 questionnaire, scores were transformed into 0 to 100 scales, with a score of 0 represented the worst possible health-related quality of life and a score of 100 representing the most favorable health-related quality of life. The questionnaire will be administered once; 12 months after the patient's initial consultation.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care)
Number analyzed (Participants) | 5 | 6 | 7
score on a scale
  Urinary Incontinence: number analyzed (Participants) | 5 | 4 | 7
  Urinary Incontinence | 79.7 [58.5 to 100] | 67.2 [16.5 to 93.8] | 85.8 [60.5 to 100]
  Urinary Irritative: number analyzed (Participants) | 5 | 5 | 7
  Urinary Irritative | 80.0 [43.8 to 93.8] | 90.0 [81.2 to 100] | 83.9 [56.2 to 100]
  Bowel | 86.7 [62.5 to 100] | 72.9 [29.2 to 100] | 92.3 [58.3 to 100]
  Sexual: number analyzed (Participants) | 5 | 4 | 7
  Sexual | 29.4 [0 to 70.8] | 35.1 [12.5 to 73.7] | 20.2 [16.7 to 27.8]
  Hormonal: number analyzed (Participants) | 5 | 5 | 7
  Hormonal | 86.0 [60.0 to 100] | 80.0 [60 to 95] | 76.4 [60 to 100]

4. Secondary Outcome: Utilization as Determined by Chart Review
Description: Will be categorized by the type of treatment the patient elected to receive. Will be compared across intervention arms.
Time Frame: 12 months
Population: Secondary outcomes were to be based on data collected at 12 months. Treatment choice could be ascertained immediately upon patient treatment selection. Two of our sites (enrolling >50% of study participants) experienced staff turnover and/or loss of contact with participants. As a result, we lost our ability and opportunity to maintain contact with several participants and were unable to collect treatment choice for all participants. Results reported reflect the data we were able to collect.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care)
Number analyzed (Participants) | 26 | 21 | 24
Participants
  Radical prostatectomy | 1 | 0 | 1
  Laparoscopic radical prostatectomy | 0 | 0 | 0
  Robotic-assisted laparoscopic radical prostatectomy | 14 | 14 | 12
  Cryosurgery | 0 | 0 | 0
  Intensity modulated radiation therapy (IMRT) | 3 | 6 | 8
  Brachytherapy | 4 | 0 | 2
  Proton beam | 1 | 0 | 1
  Hormone therapy | 4 | 4 | 10
  Chemotherapy | 0 | 0 | 0
  Active surveillance | 3 | 2 | 1

ADVERSE EVENTS:
Description: This study did not collect adverse events.
  We do not anticipate any additional adverse events related to participation in this study beyond usual care. If patients experience any emotional discomfort when completing the questionnaires, they may choose not to complete them and/or speak with the site staff. Patients experiencing any physical or psychological complications related to their standard of care treatment should discuss this with their treating physician.
Arm/Group | Arm A (Knowing Your Options) | Arm B (Prostate Choice) | Arm C (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT03182998/Prot_SAP_000.pdf